CLINICAL TRIAL: NCT04571606
Title: Interscalene Catheter vs. Interscalene Liposomal Bupivacaine for Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-3303
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): Pre-operative ultrasound guided interscalene nerve block with 10 mL 1.3% liposomal bupivacaine (Exparel) and 10 mL 0.5% bupivacaine
  Interventions: Procedure: Single injection peripheral nerve block with liposomal bupivacaine (Exparel)
- Peripheral Nerve Catheter (Active Comparator): Pre-operative ultrasound guided interscalene nerve block with 20 mL of 0.25% bupivacaine and placement of peripheral nerve catheter with 10 mL/hr 0.2% bupivacaine infusion via OnQ pump.
  Interventions: Procedure: Single injection peripheral nerve block with 0.25% bupivacaine and subsequent peripheral nerve catheter with 0.2% bupivacaine infusion via onQ pain pump

INTERVENTIONS:
Procedure: Single injection peripheral nerve block with liposomal bupivacaine (Exparel) — 10 mL/133 mg liposomal bupivacaine and 10 mL 0.5% bupivacaine
  Arms: Liposomal Bupivacaine
Procedure: Single injection peripheral nerve block with 0.25% bupivacaine and subsequent peripheral nerve catheter with 0.2% bupivacaine infusion via onQ pain pump — 20 mL 0.25% bupivacaine block and subsequent 10 mL/hr 0.2% bupivacaine infusion for 48 hours
  Arms: Peripheral Nerve Catheter

SUMMARY:
Arthroscopic rotator cuff repair often causes significant postoperative pain. An interscalene nerve catheter is an effective and proven method to help reduce postoperative pain and decrease opioid use around the time of shoulder surgery. Liposomal bupivacaine (Exparel) was recently approved by the FDA for use around the interscalene brachial plexus, and it has been shown to be an effective option, but its analgesic efficacy has limited data. Both techniques are currently being used at the UNC's Ambulatory Surgery Center (ASC) for analgesia after shoulder arthroscopy. The goal is to ensure that the fairly new Exparel option provides non-inferior analgesia as compared to the prior standard practice of placing a nerve catheter with plain bupivacaine. The investigators hope to ensure the quality of pain control around the time of shoulder arthroscopy at this institution by prospectively and rigorously collecting data during regular follow up.

DETAILED DESCRIPTION:
This is a prospective comparison of patients undergoing rotator cuff repair that receive one of two types of interscalene nerve block, both of which are currently being used at UNC. Group 1 will be comprised of patients with a preoperative interscalene nerve catheter placed with 20 mL 0.25% bupivacaine and a 0.2% ropivacaine infusion by an OnQ pain pump. Group 2 will be comprised of patients with a preoperative interscalene nerve block placed with 10 mL 0.5% bupivacaine and 10 mL 1.3% Liposomal Bupivacaine (Exparel). All patients in both groups will have a similar intraoperative general anesthetic with multimodal analgesic pre-op oral medications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age > 18 undergoing arthroscopic rotator cuff repair at the ambulatory surgery center at the University of North Carolina

Exclusion Criteria: the below are simply contraindications to regional anesthesia in general, this is a pragmatic study to evaluate the quality of care for these patients with no additional exclusion criteria.

* Contraindications to regional anesthesia
* Significant peripheral neuropathy or neurological disorder affecting the upper extremity
* Pregnancy
* Cognitive or psychiatric condition that might affect patient assessment and/or inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 15 Score (QOR15) | 48 hours postoperatively
  The QoR15 provides a valid, extensive, and efficient evaluation of postoperative quality of recovery. The QOR15 has 15 questions on a 0-10 point scale, so the QOR15 score can range from 0-150, the higher the score, the better the quality of recovery.

OTHER OUTCOMES:
Opioid Dose in Morphine Equivalents | postoperative days 1, 2 & 3
  total opioid administered over the first 3 postoperative days
Percentage of Patients with a Highest Pain Score > 3 | postoperative days 1, 2 & 3
  Visual analog pain scores after operation [0-10, with 10 being the worst pain]

CONTACTS AND LOCATIONS:
Overall Officials: Jay Schoenherr, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Ambulatory Surgery Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC